CLINICAL TRIAL: NCT02050451
Title: A Pilot Study of Perioperative Oral Nutrition Supplementation to Improve Nutritional Status, Post-operative Complications, Length of Stay and Readmission Rates in Patients Undergoing Radical Cystectomy
Brief Title: Perioperative Oral Nutrition Intervention for Patients Undergoing Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Chad Ritch, Clinical Instructor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VU-IRB-131560
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Bladder Cancer
Keywords: radical cystectomy; urinary diversion; nutrition; oral supplementation; enteral nutrition
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Ensure Plus; Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition Intervention (Experimental): Ensure Plus®, consumed orally twice daily for 2 weeks before and 4 weeks after surgery
  Interventions: Dietary Supplement: Ensure Plus®
- Control (Active Comparator): Over the counter daily multivitamin for 2 weeks before and 4 weeks after surgery
  Interventions: Dietary Supplement: Multivitamin

INTERVENTIONS:
Dietary Supplement: Ensure Plus®
  Other Names: Ensure®
  Arms: Nutrition Intervention
Dietary Supplement: Multivitamin
  Arms: Control

SUMMARY:
The current study is designed to assess the impact of an enriched oral nutritional shake (Ensure Plus®) to improve the nutritional status and patient outcome after surgery to remove a cancerous bladder (radical cystectomy). Radical cystectomy with urinary diversion using a segment of intestine is the standard of care for invasive bladder cancer. This operation has a high complication rate and several studies have shown that this may be directly related to poor nutrition.

The investigators believe that patients who consume an enriched nutritional shake before and after surgery will improve their nutrition status and experience fewer complications, shorter length of stay and less readmissions compared to those who do not.

Patients who are scheduled to undergo elective radical cystectomy will be eligible for enrollment. Once enrolled, they will be randomly assigned to one of two groups. One group will be offered Ensure Plus® twice daily for 2 weeks before and 4 weeks after their surgery and the other will be offered a daily over-the-counter multivitamin for the same period of time. The investigators will follow both groups for up to 30 days after their surgery and compare clinical outcomes such as: complication rates, length of stay, readmission rates and mortality as well as measure serum markers of nutrition status and assess changes in body composition.

ELIGIBILITY:
Inclusion Criteria:

* all patients eligible for elective radical cystectomy for bladder cancer at the sponsoring institution

Exclusion Criteria:

* inability to tolerate oral supplementation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Hospital-free days (HFDs) | 30 days
  The study is powered to detect a difference in the number of HFDs over a 30 day period between intervention and control groups

SECONDARY OUTCOMES:
Serum markers | 30 days
  The investigators will compare serum levels of albumin, prealbumin, transferrin and retinol binding protein and C-reactive protein between groups
Body composition | 30 days
  The investigators will measure difference in lean body mass and fat mass between intervention and controls using whole body dual energy X-ray absorptiometry (DEXA) scan
Tolerability / compliance | 30 days
  The investigators will assess the patients' ability to tolerate and comply with the nutrition intervention
Complications | 30 days
  The investigators will compare the difference in rate, type and severity of post-operative complications between groups
Length of stay | 30 days
  The investigators will compare the length of stay following surgery between the two groups
Readmission rate | 30 days
  The investigators will compare the rate of readmissions over the 30 day postoperative period between intervention and control
Mortality | 30 days
  The investigators will compare overall survival between groups over the 30 day postoperative period
Calories | 30 days
  The investigators will compare caloric and nutrient intake between groups using comprehensive dietary assessment tools

CONTACTS AND LOCATIONS:
Overall Officials: Chad R Ritch, MD, Principal Investigator — Department of Urologic Surgery, Vanderbilt University Medical Center; Michael S Cookson, MD, Study Director — Department of Urology, University of Oklahoma Medical Center; Heidi J Silver, PhD, RD, Study Director — Vanderbilt Center for Human Nutrition; Peter E Clark, MD, Study Director — Department of Urologic Surgery, Vanderbilt University Medical Center; Sam S Chang, MD, Study Director — Department of Urologic Surgery, Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Gregg JR, Cookson MS, Phillips S, Salem S, Chang SS, Clark PE, Davis R, Stimson CJ Jr, Aghazadeh M, Smith JA Jr, Barocas DA. Effect of preoperative nutritional deficiency on mortality after radical cystectomy for bladder cancer. J Urol. 2011 Jan;185(1):90-6. doi: 10.1016/j.juro.2010.09.021. Epub 2010 Nov 12. PMID 21074802
- [Background] Stimson CJ, Chang SS, Barocas DA, Humphrey JE, Patel SG, Clark PE, Smith JA Jr, Cookson MS. Early and late perioperative outcomes following radical cystectomy: 90-day readmissions, morbidity and mortality in a contemporary series. J Urol. 2010 Oct;184(4):1296-300. doi: 10.1016/j.juro.2010.06.007. Epub 2010 Aug 17. PMID 20723939
- [Background] Morgan TM, Keegan KA, Barocas DA, Ruhotina N, Phillips SE, Chang SS, Penson DF, Clark PE, Smith JA Jr, Cookson MS. Predicting the probability of 90-day survival of elderly patients with bladder cancer treated with radical cystectomy. J Urol. 2011 Sep;186(3):829-34. doi: 10.1016/j.juro.2011.04.089. Epub 2011 Jul 23. PMID 21788035